CLINICAL TRIAL: NCT01513980
Title: RENEWING HEALTH - Large Scale Pilot in Veneto Region: Life-long Monitoring in COPD
Brief Title: Life-long Monitoring of COPD in Veneto Region
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regione Veneto (Other)
Collaborators: European Commission (Other); Azienda Unità Locale Socio Sanitaria n.9 Treviso (Other); Azienda ULSS 12 Veneziana (Other); Azienda ULSS di Verona e Provincia (Other); Azienda ULSS 16 Padova (Other); Azienda Ospedaliera di Padova (Other); Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: G. A. 250487-Veneto WP8Cl5
Record Dates: First submitted 2012-01-17; First posted 2012-01-20 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2012-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic Obstructive Pulmonary Disease; Telemonitoring
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control group (No Intervention): Treatment as usual
- Self monitoring for patients with COPD (Experimental): Procedure: self-monitoring for patients with severe COPD
  Interventions: Procedure: self-monitoring for patients with severe COPD
- Nurse monitoring for patients with COPD (Experimental): Procedure: nurse-monitoring for patients with severe COPD
  Interventions: Procedure: nurse-monitoring for patients with severe COPD

INTERVENTIONS:
Procedure: self-monitoring for patients with severe COPD — Patients are equipped with a telemonitoring kit composed by a portable wrist-clinic device for clinical parameters measuring and a gateway device for data transmission.
  The patient can monitor pulse-oxymetry and heart rate with a frequency set by the clinician in the personalised treatment plan. Data are transmitted to a regional eHealth centre where a group of operators keeps these information under control and alert the reference clinician in case of worsening of symptoms. CAT questionnaire is monthly administrated by phone to the patients
  Arms: Self monitoring for patients with COPD
Procedure: nurse-monitoring for patients with severe COPD — A nurse is in charge of data collection during home visits with a frequency set by the lung specialist depending to the patient clinical conditions. The nurse uses portable biomedical devices to measure pulse-oxymetry, heart rate, spirometry and if scheduled an arterial blood gas test. Data are transmitted to the clinician who checks them on his laptop in the hospital and completes the visit with the medical report.
  Arms: Nurse monitoring for patients with COPD

SUMMARY:
The purpose of this study is to evaluate whether the introduction of large-scale telemonitoring of patients with COPD produces benefits in terms of improved health-related quality of life and reduced access to hospital facilities. In addition, the trial evaluates the economic and organisational impact of the new services, and examine their acceptability by patients and health professionals.

DETAILED DESCRIPTION:
The study is designed to evaluate the impact of telemonitoring on the management of COPD compared with outpatient usual care. From a clinical point of view, the trial will allow to investigate how telemonitoring contributes to improve COPD patients health-related quality of life and reduct the access to hospital facilities (re-hospitalizations, bed-days, specialistic and ER visits) and the anxiety about health conditions. A cost-effectiveness and cost-utility analysis will be carried out in order to determine if and how telemonitoring helps to limit the healthcare expenditure. The evaluation will deal also with organizational changes and task shift due to telemonitoring introduction and patients and professionals perception towards the service.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* COPD GOLD class 3-4
* Life expectance > 12 months

Exclusion Criteria:

• Patient unable to use the equipment provided (alone or assisted).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Actual)
Dates: Start 2011-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Health-Related quality of life | 12 months
  Health-Related Quality of Life is assessed by the SF-36 questionnaire

SECONDARY OUTCOMES:
Number of bed days for hospitalised patients | 12 months
Number of specialist visits | 12 months
Number of visits to emergency department | 12 months
All cause mortality | 12 months
Anxiety and depression status | 12 months
  Anxiety and depression status is assessed by Hospital Anxiety and Depression Scale, (HADS).
Number of re-hospitalizations | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Fusello, MD, Principal Investigator — Local Health authority Veneziana
Locations (6):
- Italy (6):
  - Local Health Autority n.16 Padova - Pulmonology outpatient clinic, Padua, Padova
  - Hospital Trust of Padova - Respiratory Physiopathology Department, Padua, Padova
  - Ospedale Ca'Foncello - Pulmonology Department, Treviso, Treviso
  - Ospedale dell'Angelo - Pulmonology Department, Mestre, Venezia
  - Ospedale di Marzana - Rehabilitative respiratory unit, Marzana, Verona
  - Hospital Trust of Verona - Pneumonology Department, Verona, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vianello A, Fusello M, Gubian L, Rinaldo C, Dario C, Concas A, Saccavini C, Battistella L, Pellizzon G, Zanardi G, Mancin S. Home telemonitoring for patients with acute exacerbation of chronic obstructive pulmonary disease: a randomized controlled trial. BMC Pulm Med. 2016 Nov 22;16(1):157. doi: 10.1186/s12890-016-0321-2. PMID 27876029
- See also: The Renewing Health project is partially funded under the ICT Policy Support Programme (ICT PSP) as part of the Competitiveness and Innovation Framework Programme by the European Community — http://www.renewinghealth.eu